CLINICAL TRIAL: NCT04906161
Title: Correlation Between Vitamin D and Serum Calcium Level Insufficiency and Early Dental Implant Failure
Brief Title: Vitamin D and Serum Calcium Level Insufficiency and Early Dental Implant Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Doaa Adel Salah Khattab, Principle investigator, Ain Shams University
Other Study IDs: 1388
Record Dates: First submitted 2021-05-06; First posted 2021-05-28 (Actual); Last update posted 2021-05-28 (Actual); Status verified 2021-05

CONDITIONS: Vitamin D Deficiency; Dental Implant Failure Nos
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Successful dental implant: Patients showed a successful implant placement with no complications before loading
  Interventions: Diagnostic Test: Vitamin D and calcium levels
- Early dental implant failure: Early complications and failure of dental implant before loading
  Interventions: Diagnostic Test: Vitamin D and calcium levels

INTERVENTIONS:
Diagnostic Test: Vitamin D and calcium levels — Mini VIDAS® compact multiparametric immunoanalyzer for vitamin D analysis (BIOMERIEUX- France)

SUMMARY:
In this study there is a trial to investigate whether there is a correlation between early implant failure and low serum levels of vitamin D.

DETAILED DESCRIPTION:
Osseointegration is a complex phenomenon and depends on many factors; some are related to the implant (material, macroscopic design, and implant surface), others to the surgical-prosthetic protocol (surgical technique, loading conditions, and time), and others to the patient (quantity/quality of bone at the receiving site and the host response)

All these observations would suggest the existence of specific patient-related risk factors such as vitamin D deficiency in the blood, could play an important role in the occurrence of early dental implant failures (EDIFs), but unfortunately are neglected by the dental literature.

In this study there is a trial to investigate whether there is a correlation between early implant failure and low serum levels of vitamin D. Therefore we are including patients with early implant failure during the year 2020 using the same implant (material, macroscopic design, and implant surface), surgical-prosthetic protocol (surgical technique, loading conditions, and time)

The study will be performed into 15 male and 15 female participants that had dental implant placement in the last 3 months. An informed consent will be signed with the patient with full detail on the study.

The situation of the implant will be categorized into either successful or failed dental implant.

Medical history and lifestyle information will be obtained by questionnaire. Levels of serum vitamin D will be collected from participants

Statistical analysis will correlate between vitamin D and early implant failure.

ELIGIBILITY:
Inclusion Criteria:

* Missing single tooth
* Systemically free
* Average body mass index

Exclusion Criteria:

* Systemic conditions
* Bad oral hygiene

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Multicenter study on systemically free participants that had a dental implant within the last 6 months using the same implant system, preoperative planning techniques, surgical protocol (minimal invasive implant concept), post surgical protocol and excluding any cases with intrasurgical difficulties and complications.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-07-20 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Implant success with normal serum vitamin D level | 6 months
  Implant stability with no further radiographic bone loss following bone remodeling with successful prosthetic part
Early implant failure with deficient serum vitamin D level | 6 months
  Mobile extruded implant with radiographic bone loss and peri-implant pathosis

CONTACTS AND LOCATIONS:
Overall Officials: Bassem E Abd ElMoneim Hussein, MDs, Principal Investigator — Ain Shams University
Locations (2):
- Egypt (2):
  - Ain Shams University, Cairo, Abbassia
  - Doaa Khattab, Cairo, Abbassia

IPD SHARING:
Plan to Share IPD: No